Participant ID Number: \_\_\_ (for researcher use)

## PARTICIPANT CONSENT FORM

## Does Sound Conditioning Protect Against Temporary Hearing Damage?

Name of Co-Investigator: Hemna Santilale

Chief Investigator: Emily Frost

Academic Supervisor: Prof. Chris Plack, University of Manchester

| | | Please initial | each box |
|---|---|---|---|
| 1. I confirm that I have read and understand the subject information sheet dated 21/01/2019 Version 4 for the above study and have had the opportunity to ask questions which have been answered fully. | | | |
| 2. I understand that my participation is voluntary and I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. I understand that sections of any of my research notes may be looked at by responsible individuals from Imperial College Healthcare NHS Trust or from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to access my records that are relevant to this research. | | | |
| 4. Where any tests may indicate an abnormal result, I agree that a letter will be sent to my GP with a copy of all test results. | | | |
| 5. I understand that the interview will be recorded. I give permission for this recording to take place. I understand that this recording will be deleted or destroyed once it has been transcribed. | | | |
| 6. I agree to take part in the above study. | | | |
| Name of Patient/Participant | Signature | Date | |
| Hemna Santilale Principal Investigator | Signature | | |